CLINICAL TRIAL: NCT07348601
Title: A Proof-of-Concept Open-Label Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of CSTI-500 in Participants With Prader-Willi Syndrome
Brief Title: A Study of CSTI-500 in Patients With Prader-Willi Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ConSynance Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CSTI-500-005
Record Dates: First submitted 2025-12-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prader-Willi Syndrome
Keywords: PWS; Prader-Willi Syndrome; CSTI-500
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CSTI-500 (Open-label) Low Target Exposure (Experimental)
  Interventions: Drug: CSTI-500
- CSTI-500 (Open-Label) Medium Target Exposure (Experimental)
  Interventions: Drug: CSTI-500
- CSTI-500 (Open-label) High Target Exposure (Experimental)
  Interventions: Drug: CSTI-500

INTERVENTIONS:
Drug: CSTI-500 — CSTI-500 given orally in an open-label, dose-escalation design with individualized dosing.

SUMMARY:
This is a proof-of-concept, open-label, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of CSTI-500 in participants with genetically confirmed Prader-Willi Syndrome (PWS) who are 13 to 50 years of age. Participants will receive increasing doses of CSTI-500, and blood levels will be measured to guide individualized dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male and female individuals between the ages of 13 and 50, inclusive
2. Documented medical record history of PWS confirmed by genetic testing and PWS Nutritional Phase 3
3. CGI-S score ≥4 at Screening and Baseline (behavioral)
4. Screening HQ CT total scores ≥ 13
5. Participants must not be taking SSRI, SNRI, DNRI (bupropion), tricyclic antidepressants, stimulants, antipsychotic medications, and MAO inhibitors within 30 days of screening and willing to not start taking these medications while on the study. Fluoxetine is exclusionary unless treatment has been discontinued >6 months prior to Screening.
6. Caregiver/parent must agree to bring the subject to the site for the visits, remain with the subject during visit times when allowed and respond to any questions.
7. Caregiver/parent is willing to provide informed consent and agrees to adhere to required study procedures including telemedicine visits, visit duration requirements, and offer consistent care.
8. Caregivers must agree to complete all study required assessments.
9. Participants who cannot consent for themselves and are able will provide assent.
10. Female participants must not be pregnant or lactating. Nonpregnancy will be confirmed for all females by a urine pregnancy test conducted at Screening and at the Baseline Visit prior to enrollment into the study. If of childbearing potential, the subject/caregiver agrees to the use of one of the accepted contraceptive regimens from Screening to the first administration of the study medication, during the study, and for at least 30 days after the last dose of the study medication. An acceptable method of contraception includes one of the following:

    1. Hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
    2. Intrauterine device (with or without hormones)
    3. OR agrees to use a double barrier method (e.g., condom and spermicide) during the study and for at least 30 days after the last dose of the study medication.
    4. The investigator can use their judgement and familiarity with the participant's preferred and usual lifestyle to understand which form of birth control would be the best and also to determine if abstinence is an option that would achieve 100% effectiveness.
11. If the female is of non-childbearing potential -surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is postmenopausal (at least 1 year without menses) as confirmed by follicle-stimulating hormone (FSH) levels of ≥ 40 mIU/mL. No contraceptive use is required.
12. Unless, sterile, a male study subject/caregiver must agree to use a double barrier method (e.g., condom and spermicide).
13. For adults, supine systolic blood pressure must be ≤140 mmHg and ≥100 mmHg; diastolic blood pressure must be ≤80 mmHg and ≥60 mmHg at Screening. Heart rate must be ≥50 bpm and ≤100 bpm. Heart rate increase on standing must be within acceptable range (see exclusion criterion 10).

    For adolescents, a systolic and diastolic BP that is between the 5th and 90th percentile for age and sex.

    a. Two repeat measurements within 10 minutes of the first reading are permitted at the discretion of the Investigator. If this option is used, the last obtained reading will be used for determination of eligibility. Averages will not be used.
14. All concomitant medications including blood pressure medications and type 2 diabetic medications must be stable for ≥3 months prior to screening (≤10% change) and there must be no medication changes (dose change, initiation, discontinuation) intentionally planned during the study. Supplements and vitamins are not considered concomitant medications for eligibility purposes.
15. Stated willingness to comply with all study procedures including visits, restrictions, and availability for the duration of the study.

Exclusion Criteria:

1. Participation in any clinical study with an investigational drug/device within 3 months prior to screening or during the study
2. PWS diagnosis of UPD (maternal uniparental disomy).
3. Current use of DCCR or if used previously, must be off at least 4 weeks before screening.
4. Recent use (within 3 months) of weight loss agents including prescription, herbal medications, and weight loss supplements. Ozempic, for diabetes, would be exclusionary due to its effect on weight loss.
5. History of bariatric surgery or major surgery within 6 months of screening or planned during the study.
6. Any malignancy in the 2 years prior to screening (excluding basal cell carcinoma or squamous cell carcinoma of the skin or cervical carcinoma in situ that have been successfully treated).
7. Current liver, pulmonary, cardiac, or GI disease that would be expected to adversely affect study participation. Stable disease, e.g., asthma or controlled hypertension is not excluded. Liver disease or liver injury as indicated by abnormal liver function tests, ALT, AST, alkaline phosphatase, or serum bilirubin (≥3X ULN for any of these tests).

   a. Participants with impaired liver function (Child-Pugh Scores A, B, C)
8. Unexplained history or presence of combination of unexplained symptoms e.g., dizziness, syncope, fatigue, palpitations/tachycardia, headaches, or exercise intolerance.
9. Prohibited Medications include SSRI, SNRI, DNRI (bupropion), tricyclic antidepressants, stimulants, antipsychotics, MAO inhibitors, fluoxetine, mood stabilizers, and GLP-1 agonists
10. Presence of postural orthostatic tachycardia syndrome (POTS) for any reason, defined as:

    1. For participants aged 19 or older, sustained heart rate increase of >30 bpm or an increase to 120 bpm or greater within 3 minutes of standing.
    2. For participants aged 13-19, a sustained heart rate increase of >40 bpm or an increase to 120 bpm or greater within 3 minutes of standing.
    3. Associated with related symptoms that are worse with upright posture and that improve with recumbence.
11. A clinically significant abnormal finding on 12-lead electrocardiogram (ECG) at Screening. Note QT corrected according to Fridericia's formula (QTcF) interval of ≥450 msec will be exclusionary [QTc = QT/(RR^0.33)]. The ECG may be repeated once for confirmatory purposes if initial values obtained exceed the limits specified.
12. Any clinically significant cardiac arrhythmia (e.g., atrial fibrillation, Adams-Stokes's disease, Wolff-Parkinson-White syndrome, atrioventricular block 2nd or 3rd degree).
13. Heart failure classified per the New York Heart Association (NYHA) as level II or greater.
14. Myocardial infarction, stroke, or confirmed TIA within the last 5 years.
15. Estimated glomerular filtration rate (eGFR) ≤ 90 mL/min/1.73m² for ages 13 to <18 years of age. For adults ≥18 years of age, body-surface area corrected eGFR and exclusion with eGFR <90 mL/min.
16. Uncontrolled Type 2 diabetes as defined by HbA1c ≥ 9% at Screening.
17. Insulin-dependent Type 1 diabetes.
18. Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies with detected circulating ribonucleic acid (RNA), or HIV 1 and 2 antibodies.
19. Uncontrolled thyroid disease.
20. Known hypersensitivity to any component of investigational product.
21. History or active psychotic symptoms, or medical conditions which the investigator believes will interfere significantly with study compliance. Participants with a history of other severe psychiatric disorders, e.g., schizophrenia, major depressive disorder, bipolar disorder, or other DSM-V disorders.
22. History of any suicidal behavior.
23. Known alcohol or substance abuse.
24. Moderate to strong inhibitors/inducers of CYP2D6, CYP3A4 and CYP2C9, including grapefruit juice. Substrates of CYP1A2 and CYP2B6.
25. Any other medical, physical, or personal issues which, in the opinion of the investigator, would interfere with the subject's ability to complete the trial per protocol.
26. Inability to swallow the oral capsules whole with water.

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 14 weeks
  Number of participants with TEAEs, defined as an adverse event (AE) that is new or worsened in severity after the dose of study drug (coded using MedDRA).
Proportion achieving target CSTI-500 steady-state Cmax with PK-guided dose individualization | 12 weeks
  Proportion of participants whose observed CSTI-500 steady-state Cmax is within the protocol-defined target range for the assigned target concentration level, using plasma concentrations measured from scheduled PK sampling to guide dose adjustments.
Incidence of clinically significant findings in laboratory values | 12 weeks
  Laboratory evaluations include hematology, blood chemistry, and urinalysis parameters.
Incidence of clinically significant findings in 12-lead electrocardiograms (ECGs) | 12 weeks
  QT interval, corrected QT interval (QTc), PR interval, QRS duration, and heart rate will be measured by 12-lead electrocardiogram.
Incidence of clinically significant findings in vital signs | 12 weeks
  Participants will be assessed for any clinically significant changes in vital parameters (systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate, and body temperature).

SECONDARY OUTCOMES:
Change from baseline in Hyperphagia Questionnaire for Clinical Trials (HQ-CT) total score | 12 weeks
  Change from baseline in the Hyperphagia Questionnaire for Clinical Trials (HQ-CT) total score. The HQ-CT total score ranges from 0 to 36, with higher scores indicating greater hyperphagia.
Change from baseline in Aberrant Behavior Checklist - Community (ABC-C) total score and subscale scores | 12 weeks
  Change from baseline in Aberrant Behavior Checklist - Community (ABC-C) total score and subscale scores. The ABC-C is a 58-item caregiver-reported questionnaire, with higher scores indicating more severe aberrant behavior.
Clinical Global Impression-Improvement (CGI-I) score | 12 weeks
  Clinical Global Impression-Improvement (CGI-I) score assessed at Week 12. The CGI-I is a 7-point ordinal scale, with lower scores indicating greater improvement.
Change from baseline in Clinical Global Impression-Severity (CGI-S) score | 12 weeks
  Change from baseline in Clinical Global Impression-Severity (CGI-S) score. The CGI-S is a 7-point ordinal scale, with lower scores indicating less severe illness (better outcome).
Change from baseline in Prader-Willi Syndrome Questionnaire (PADQ) score | 12 weeks
  Change from baseline in the Prader-Willi Syndrome Questionnaire (PADQ) score. The PADQ is a caregiver-reported questionnaire, with higher scores indicating greater symptom severity (worse outcome).
Change from baseline in Caregiver Global Impression-Severity (careGI-S) score | 12 weeks
  Change from baseline in Caregiver Global Impression-Severity (careGI-S) score. The careGI-S is a caregiver-reported ordinal scale, with lower scores indicating less severe symptoms (better outcome).
Caregiver Global Impression-Change (careGI-C) score | 12 weeks
  Caregiver Global Impression-Change (careGI-C) score assessed at Week 12. The careGI-C is a caregiver-reported ordinal scale, with lower scores indicating greater improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No